CLINICAL TRIAL: NCT07392892
Title: A PHASE 2/3 INTERVENTIONAL STUDY OF PF-08634404 IN COMBINATION WITH CHEMOTHERAPY IN TREATMENT-NAÏVE PARTICIPANTS WITH LOCALLY ADVANCED OR METASTATIC GASTRIC, GASTROESOPHAGEAL JUNCTION, OR ESOPHAGEAL ADENOCARCINOMA
Brief Title: A Study to Learn About the Study Medicine Called PF-08634404 in Combination With Chemotherapy in Gastroesophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C6461016; 2025-524717-86-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Untreated Advanced or Metastatic Gastric, Gastroesophageal Junction , or Esophageal Adenocarcinoma; Metastatic Gastric Cancer; Gastroesophageal Junction Cancer; Esophageal Adenocarcinoma
Keywords: gastric cancer; gastroesophageal junction cancer; esophageal adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Drug Therapy; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2 is open-label, whereas Phase 3 is double-blind, randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 2 Portion (Experimental): PF-08634404 + Chemotherapy
  Interventions: Biological: PF-08634404; Drug: Chemotherapy
- Phase 3: Arm A (Experimental): PF-08634404 + Chemotherapy
  Interventions: Biological: PF-08634404; Drug: Chemotherapy
- Phase 3: Arm B (Active Comparator): Nivolumab + Chemotherapy
  Interventions: Drug: Chemotherapy; Biological: Nivolumab

INTERVENTIONS:
Biological: PF-08634404 — Participants will receive PF-08634404 intravenously.
  Other Names: SSGJ-707
  Arms: Phase 2 Portion; Phase 3: Arm A
Drug: Chemotherapy — Participants will receive PF-08634404 intravenously in combination with Chemotherapy.
Biological: Nivolumab — Participants will receive Nivolumab intravenously.
  Arms: Phase 3: Arm B

SUMMARY:
This study is being done to learn more about a new medicine called PF-08634404 and how well it works when given with chemotherapy to people with gastroesophageal cancer that is locally advanced (spread to nearby tissues) or has spread to other parts of the body.

To join the study, participants must meet the following conditions:

Be 18 years or older. Have locally advanced or metastatic gastric, gastroesophageal junction or esophageal adenocarcinoma Be treatment naïve for advanced or metastatic disease Be in good physical condition and have healthy organs based on medical tests.

The study has two parts:

* In the first part, researchers will check how safe the study medicine in combination with chemotherapy is and how well people respond to it.
* In the second part, they will compare study medicine plus chemotherapy to another approved treatment (nivolumab plus chemotherapy) to see which works better.

The treatment will be given in repeated time periods called cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed gastric, gastroesophageal junction or esophageal adenocarcinoma.
* Evidence of locally advanced or metastatic disease.
* Eastern Cooperative Oncology Group performance status (ECOG) 0-1
* No prior systemic therapy for advanced or metastatic disease.
* Adequate hepatic, liver, and renal function

Exclusion Criteria:

* Participants with known active CNS metastases, including leptomeningeal, brainstem, meningeal, or spinal cord metastases or compression
* Clinically significant risk of hemorrhage or fistula
* Major surgery or severe trauma within 4 weeks prior to the first dose, or planned major surgery during the study
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Any Grade ≥3 bleeding/hemorrhage events within 28 days of Cycle 1 Day 1, or prior history of clinically significant bleeding events
* Clinically significant cardiovascular disease, or other comorbidities, within 6 months prior to first dose
* Participants with active autoimmune diseases requiring systemic treatment within the past 2 years
* Evidence of non-infectious or drug-induced interstitial lung disease (ILD) pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2031-07-22 (Estimated); Study Completion 2032-07-21 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Confirmed Objective response rate (ORR) using RECIST 1.1 as assessed by investigator | Approximately 4 years
  Confirmed ORR by investigator is defined as the proportion of participants with confirmed Complete Response (CR) or Partial Response (PR) per RECIST v1.1 as assessed by investigator.
Phase 2: Number of participants with treatment-emergent adverse events | Through 90 days after the last study intervention; Approximately 4 years
  Adverse Events (AEs) as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study intervention.
Phase 3: Progression Free Survival (PFS) using RECIST 1.1 as assessed by BICR | Approximately 4 years
  PFS by BICR is defined as the time from the date of randomization to the date of first documented disease progression per RECIST 1.1 as assessed by BICR, or death due to any cause, whichever occurs first.
Phase 3: Overall Survival (OS) | Approximately 4 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Phase 2: Duration of Response (DOR) using RECIST 1.1 as assessed by investigator | Approximately 4 years
  DOR by investigator is defined as the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, respectively, or death due to any cause, whichever occurs first.
Phase 2: Progression Free Survival (PFS) using RECIST 1.1 as assessed by investigator | Approximately 4 years
  PFS by investigator is defined as the time from the date of first dose to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, or death due to any cause, whichever occurs first.
Phase 2: Overall Survival (OS) | Approximately 4 years
  OS is defined as the time from the date of first dose to the date of death due to any cause.
Phase 2: Number of participants with laboratory abnormalities | Through 90 days after the last study intervention; Approximately 4 years
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, high, low, or not done and be listed.
Phase 2: Serum concentrations of PF-08634404 | Approximately 21 months
  Predose and postdose concentrations of PF-08634404
Phase 2: Incidence of Anti-Drug Antibody (ADA) against PF-08634404 | Approximately 21 months
Phase 3: ORR using RECIST 1.1 as assessed by BICR | Approximately 4 years
  ORR by BICR is defined as the proportion of participants with a Best Overall Response (BOR) of confirmed CR or confirmed PR per RECIST 1.1 as assessed by BICR.
Phase 3: ORR using RECIST 1.1 as assessed by investigator | Approximately 4 years
  ORR by investigator is defined as the proportion of participants with a BOR of confirmed CR or confirmed PR per RECIST 1.1 as assessed by investigator.
Phase 3: Progression free survival (PFS) using RECIST 1.1 as assessed by investigator | Approximately 4 years
  PFS by investigator is defined as the time from the date of randomization to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, or death due to any cause, whichever occurs first
Phase 3: DOR using RECIST 1.1 as assessed by BICR | Approximately 4 years
  DOR is defined as the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST 1.1 as assessed by BICR, respectively, or death due to any cause, whichever occurs first.
Phase 3: DOR using RECIST 1.1 as assessed by investigator | Approximately 4 years
  DOR is defined as the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, respectively, or death due to any cause, whichever occurs first.
Phase 3: PFS2 (PFS after next-line therapy) by investigator | Approximately 4 years
  PFS2 is defined as the time from the date of randomization to the date of second objective disease progression or death due to any cause, whichever occurs first
Phase 3: Number of participants with treatment-emergent adverse events | Through 90 days after the last study intervention; Approximately 4 years
  AEs as characterized by type, frequency, intensity as graded by NCI CTCAE version 5.0, timing, seriousness, and relationship to study intervention(s)
Phase 3: Number of participants with laboratory abnormalities | Through 90 days after the last study intervention; Approximately 4 years
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, high, low, or not done and be listed.
Phase 3: Serum concentrations of PF-08634404 | Approximately 21 months
  Predose and postdose concentrations of PF-08634404
Phase 3: Incidence of ADA against PF-08634404 | Approximately 21 months
Phase 3: Change from baseline in Functional Assessment of Cancer Therapy - Gastric (FACT-Ga) Total score | Approximately 4 years
Phase 3: Time to definitive deterioration in FACT-Ga Total score | Approximately 4 years
Phase 3: Time to definitive deterioration in Gastric Cancer Subscale (GaCS) score | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests